CLINICAL TRIAL: NCT00242645
Title: Computer-Assisted Cancer Risk Behavior Counseling
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively terminated.
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04F.244; K07-CA91976-0; K07CA091976 (NIH)
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes; Diabetes Mellitus; Hypertension
Keywords: Doctor-Patient relation; Physician-Patient relation; Diabetes; Office visits; Comparative Study; Health behavior; Randomized controlled trials; Health Promotion; Health Education; Computer-tailor information
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Health Behavior; Health Education | interventions — Preventive Health Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Health Information
Behavioral: Preventive Services
Behavioral: Computer tailored information

SUMMARY:
To test whether or not giving patients information before their doctor visits changes the care they receive and what type of information is best to give before the doctor visit.

DETAILED DESCRIPTION:
Patients are randomized into one of three groups. Before a single visit with diabetes care provider, the patient is called to answer interview questions about their health, diabetic care and behavior habits. After a patient visits with their doctor, they are called again to answer question about the visit they just had. If a patient is place into group A or B, based on their answers to the questions they are mailed a printed report before their doctor visit. The report will indicate how things are going the patient's diabetic care and recommended questions to ask his/her health care provided about diabetes. Group A feedback report will emphasize the risks from diabetes and the feedback reports for Group B will emphasize things to do to protect oneself from problems from having diabetes. Participants randomized to Group C will only receive printed reports after a doctors visit. No extra visit will be scheduled with the participants doctor, no travel is required, no blood tests are required and ther doctor will not be involved in the study unless the study participant chooses to discuss it with his/her doctor.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Has type 2 (adult-onset) diabetes;
* Developed diabetes after the age of 21;
* Has a scheduled doctor visit about diabetes in the next few months

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To test the effect of receiving computer tailored information about diabetes care before doctor visits and the differential effect of varying types of information

SECONDARY OUTCOMES:
Patient exit interviews after doctor visits about what happened during the visits, such as what was discussed, what tests and consults were ordered and what medications were added or changed.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N Sciamanna, MD, Study Chair — Thomas Jefferson Unversity